CLINICAL TRIAL: NCT02191540
Title: A Phase 3, Multi-Center, Single-Arm, Open-Label Study For The Safety And Efficacy Of Mistletoe Extract (AbnobaViscum® Injection) In Malignant Pleural Effusions
Brief Title: Efficacy and Safety Study of Abnoba Viscum F 20mg in Malignant Pleural Effusion Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abnoba Korea (Industry)
Collaborators: Abnoba Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-MPE-2010
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — viscum album peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abnoba Viscum F 20mg (Experimental)
  Interventions: Drug: Abnoba Viscum F 20mg

INTERVENTIONS:
Drug: Abnoba Viscum F 20mg — intravesical instillation of five amples of AbnobaViscum® F20mg and 0.9% normal saline into the pleural space
  Other Names: viscum album extract; mistletoe extract; abnobaVISCUM

SUMMARY:
Phase 3, non-randomized, Multicenter, single arm study to assess efficacy and safety of Abnoba viscum F 20mg in patients with malignant pleural effusion

ELIGIBILITY:
Inclusion Criteria:

* Subject who need the pleurodesis among subjects diagnosed with a mlignant pleural effusion
* Full lung expansion must be achieved within 12 to 24 hours after drainage
* Expected survival time of at least 2 months
* Subject who score 50 or more on the Karnofsky Performance Scale

Exclusion Criteria:

* Subjects with previous attempts at pleurodesis with sclerosing agent
* Subjects with trapped lung or bronchial obstruction
* Subjects with adverse drug response to mistletoe agents
* Subjects who have participated in another clinical study other than the present study
* Subjects who is taking immune-suppressive agents
* Subjects with medical and psychiatric contraindications for the study drug
* Subjects who are not allowed to participate in the study by legal requirement
* Subjects who are not allowed to participate in the study by the Investigator's discretion

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | 4 weeks
  Efficacy assessment of pleural effusion with Chest X-ray after 4 weeks of final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kook Joo Na, MD, Principal Investigator — Chonnam National University Hospital; Friedemann Schad, MD, Principal Investigator — FORSCHUNGSINSTITUT HAVELHOHE; YongJik Lee, MD, Principal Investigator — Ulsan University Hospital; Yeong Dae Kim, MD, Principal Investigator — Busan University Hospital
Locations (3):
- South Korea (3):
  - Busan University Hospital, Busan, Busan
  - Chonnam National University Hwasun hospital, Hwasun Gun, Jeollanam-do
  - Ulsan University Hospital, Ulsan, Ulsan